CLINICAL TRIAL: NCT01025479
Title: Prevalence of Osteoporosis in Korean Prostate Cancer Patients Who is Receiving LHRH Agonist and/or Anti-androgen Agent
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: AstraZeneca, AstraZeneca MCMD
Other Study IDs: NIS-OKR-CAS-2009/1
Record Dates: First submitted 2009-12-01; First posted 2009-12-03 (Estimated); Last update posted 2010-06-30 (Estimated); Status verified 2010-06

CONDITIONS: Prostate Cancer; Osteoporosis
Keywords: Osteoporosis; Prostate cancer; LHRH agonist and/or anti-androgen agent; Korean prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms; Osteoporosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Prevalence rate of osteoporosis and it's actual management condition in Prostate cancer patients who takes LHRH antagonist and anti androgen

ELIGIBILITY:
Inclusion Criteria:

* pathologic confirmation of prostate cancer
* patients who are taking LHRH antagonist or anti- androgen or both of them within 6 months since starting.

Exclusion Criteria:

* patients who are hard to be analysed by limitation of chart record according to investigators'discretion
* patients who already have been registered in this study

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Korean prostate cancer patients who are taking LHRH antagonist or anti- androgen or both of them within 6 months since starting.
Sampling Method: Probability Sample
Enrollment: 829 (Actual)
Dates: Start 2009-11; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
To define prevalence rate of osteoporosis in Prostate cancer patients who take LHRH antagonist or anti androgen (include MAB) at the stage of before treatment or it's initial stage.

SECONDARY OUTCOMES:
To assess whether proper osteoporosis prevention and treatment was given or not according to osteoporosis treatment guideline in prostate cancer patients who are enrolled in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Joon Woo Bahn, MD, Study Director — AstraZeneca Korea
Locations (18):
- South Korea (18):
  - Research Site, Cheonan-si, Chungcheongnam-do
  - Research Site, Gangneung-si, Gangwon-do
  - Research Site, Goyang-si, Gyeonggi-do
  - Research Site, Guri-si, Gyeonggi-do
  - Research Site, Gumi, Gyeongsangbuk-do
  - Research Site, Gyeongju, Gyeongsangbuk-do
  - Research Site, Masan-si, Gyeongsangnam-do
  - Research Site, Iksan-si, Jeollabuk-do
  - Research Site, Cheongju-si, North Chungcheong
  - Research Site, Chungju, North Chungcheong
  - Research Site, Daegu
  - Research Site, Daejeon
  - Research Site, Gwangju
  - Research Site, Incheon
  - Research Site, Jeju City
  - Research Site, Pusan
  - Research Site, Seoul
  - Research Site, Ulsan